CLINICAL TRIAL: NCT02458911
Title: Luminor Registry: Registry of the Results of Angioplasty With Drug-eluting Balloon (Paclitaxel) in the Treatment of Infrainguinal Occlusive Lesions (Superficial Femoral Artery (SFA), Popliteal Artery (PA) and Tibial Arteries (ATs)) and Restenosis From Prior Endovascular Procedures in This Sector.
Brief Title: Luminor Registry: Registry of the Results of Angioplasty With Drug-eluting Balloon (Paclitaxel) in the Treatment of Infrainguinal Occlusive Lesions and Restenosis From Prior Endovascular Procedures in This Sector.
Status: Completed | Type: Observational
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: Luminor
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Paclitaxel-eluting balloon
  Other Names: Luminor 14 & Luminor 35

SUMMARY:
The purpose of the study is to obtain data regarding safety and efficacy of drug-eluting balloon luminor 14 & luminor 35 in the treatment of infrainguinal occlusive lesions (superficial femoral artery (SFA), popliteal artery (PA) and tibial arteries (ATs)) and restenosis from prior endovascular procedures in this sector.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged at least 18
* Primary injuries and restenosis of the infrainguinal sector of AFS, AP and ATs, and intrastent restenosis or post-ATP prior in that sector.

  * Stenosis >50% and occlusions. (image test)
  * Length: 20 to 200 mm
  * Artery diameter: 2-7 mm.
* Symptomatic patients (grades 2-5 Rutherford-Baker both included; Fontaine II-IV), affected in their quality of life and that accept treatment (moderate / severe claudication patients, critical ischemia without gangrene or injuries severe enough to foresee limb amputation).

Exclusion Criteria:

* Patients with acute or subacute ischemia will be excluded.
* Existence of flow-limiting lesions in arteries of the "in flow" or the "out flow" of the sector or artery under treatment (> 50 % of the arterial diameter).
* Aneurysmal dilatation in the ipsilateral arterial axis.
* Intolerance / allergy to heparin, thienopyridine derivatives (clopidogrel , ticlopidine) and aspirin.
* Hemorrhagic diathesis during the 3 months prior to inclusion.
* Patients with a life expectancy of less than 12 months.
* Serious allergy to contrasts or PTX.
* Inability to cross the lesion with the guide (these cases will be recorded for the analysis as "intention to treat).
* Those participating simultaneously in another clinical trial.
* Pregnancy or lactation (pregnancy tests on fertiles).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery disease due to occlusive lesions, stenosis of ingraguinal arteries and restenosis after previous angioplasty with/without stent in that sector
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2014-05; Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Primary patency | 1 year
  Primary patency (performance target) of the angioplasty (PTA) performed with drug eluting balloons (DEB) in stenotic/occlusive primary lesions, in restenosis of the AFS, AP and ATs, or in stents from previous procedures in these arteries, with follow-up of 12 months.
Freedom of adverse events | 1 year
  Freedom of adverse effects (AE). EA are considered in combination: death, amputation and the need for revascularization of the target lesion (safety objective).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Getafe, Getafe, Madrid, Spain